CLINICAL TRIAL: NCT07289737
Title: Clinical Study on the Therapeutic Efficacy of Biportal Endoscopic Decompression Spine Surgery and Lumbar Decompression Fusion Surgery in the Treatment of Degenerative Lumbar Spondylolisthesis
Status: Recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2025-093
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Degenerative Spondylolisthesis
Keywords: lumbar; ube; Lumbar Degenerative Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Intraoperative resection of the ligamentum flavum, intervertebral disc, and bone tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UBE: Only decompression
- Fusion: Lumbar Spine Fusion Surgery

SUMMARY:
This study aims to systematically evaluate the therapeutic efficacy of dual-channel endoscopic spinal decompression versus lumbar decompression with fusion for degenerative lumbar spondylolisthesis. Patients undergoing either procedure will undergo detailed preoperative and postoperative follow-up to compare outcomes between the two techniques, specifically assessing postoperative pain relief, neurological improvement, and the incidence of surgical complications.

DETAILED DESCRIPTION:
1) Screening and enrollment: This study is a prospective cohort study. Patients were screened based on inclusion and exclusion criteria. They were informed that surgical treatment for degenerative lumbar spondylolisthesis could involve either lumbar fusion surgery or dual-channel endoscopic decompression alone. Specific details of both procedures were explained, allowing patients to independently choose their surgical plan. Informed consent was obtained, and baseline data including symptoms, pain scores, and neurological function scores were collected. 2) Preoperative Assessment: All patients undergo detailed pain and neurological function evaluations prior to surgery. Pain intensity is quantified using the Visual Analogue Scale (VAS), while neurological function is assessed using systems such as the JOA score and ODI score. Imaging evaluations include MRI and CT scans. 3) Data Collection: Prospective data collection was conducted for both dual-channel endoscopic spinal decompression and lumbar decompression with fusion procedures. Surgical protocols were standardized, with documentation of operative images, procedure duration, blood loss, and intraoperative complications. Spinal vertebral and accessory tissue specimens were collected during surgery. 4) Postoperative Follow-up: Patients undergo follow-up at 1 month, 3 months, 6 months, 12 months, 24 months, and 36 months postoperatively. Repeat preoperative pain and neurological function assessments, conduct regular imaging reviews, and document postoperative recovery, complication rates, and recurrence. 5) Tissue Analysis: Specimens obtained during surgery undergo histological sectioning, RT-qPCR, or Western Blot testing to analyze differences. 6) Data Analysis: Statistical software analyzes collected data to evaluate changes in pre- and postoperative pain scores, neurological function scores, and imaging outcomes. Significance testing compares the efficacy and safety of the two surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 50 and 90 years old with a confirmed diagnosis of degenerative lumbar spondylolisthesis;
2. Clinical symptoms include chronic pain, nerve compression, or motor dysfunction, confirmed by imaging studies (e.g., MRI or CT);
3. No significant improvement after at least 3 months of conservative treatment (e.g., medication, physical therapy), meeting surgical indications;
4. Understand and consent to the relevant procedures of this study, and sign the informed consent form.

Exclusion Criteria:

1. Patients exhibiting acute spinal cord compression symptoms or requiring urgent surgical intervention;
2. Patients with a history of spinal surgery or conditions such as spinal deformities, severe osteoporosis, or active infections that may compromise surgical outcomes;
3. Patients with severe comorbidities affecting assessment, such as cardiovascular disease, liver or kidney failure, or uncontrolled diabetes;
4. Patients with psychiatric disorders or cognitive impairments preventing understanding or cooperation with the study process;
5. Patients with allergies to anesthetics or surgical equipment that may increase intraoperative risks.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lumbar degenerative spondylolisthesis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
VAS | 36 month
  Pain Score
JOA score | 36month
  Function Score
ODI | 36month
  Function Score

CONTACTS AND LOCATIONS:
Locations (1):
- 4th Affiliated Hospital, School of Medicine, Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No